CLINICAL TRIAL: NCT04090970
Title: Briagen™ Case Study and Observation of Skin Excision Healing in Mohs and Other Dermatological Procedures
Brief Title: Briagen Observational Study
Acronym: BOS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gemstone Biotherapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: 1001
Record Dates: First submitted 2019-09-13; First posted 2019-09-16 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Mohs Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Briagen — Natural complex carbohydrate wound dressing for skin wounds

SUMMARY:
This research study is evaluating a study product called Briagen™ as a possible treatment for wound healing after Mohs procedure.

DETAILED DESCRIPTION:
Briagen, the study product being used in this study, is a natural complex carbohydrate wound dressing for skin wounds created by Mohs surgery.

Briagen was developed with the intent to improve healing time and reduce scarring of skin wounds. Briagen seeks to match the mechanical aspects of your skin (thickness, stiffness, hydration, pore size) to assist in the healing process.

The purpose of this research study is to observe healing time of Briagen applied to wounds created as a result of Mohs surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patient seeking treatment for wound created by Mohs or other full thickness skin excisions
2. Over 18 years of age
3. English-speaking
4. Presents for treatment within 24 hours of initial Mohs skin excision procedure.

Exclusion Criteria:

1. History of significant wound complications and non-compliance on wound maintenance instructions (infections, disturbing the wound during the healing process, etc.)
2. Known diagnosis of Diabetes
3. Active infection in the wound bed
4. Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient seeking treatment for wound created by Mohs skin excision
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-08-26 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Healing Time | 28 days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Dr. David Abramson, Englewood, New Jersey
  - Dermatology, Laser & Vein Specialists of the Carolinas, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided